CLINICAL TRIAL: NCT06160921
Title: Prognostic Model of Hypertension
Acronym: PHOP-HT
Status: Recruiting | Type: Observational
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiang Xie, Xiangxie, MD,The First Affiliated Hospital Of XinJiang Medicial University, Xinjiang Medical University
Other Study IDs: 20190818
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2
  Interventions: Other: Standard therapy

INTERVENTIONS:
Other: Standard therapy — Individualized blood pressure reduction program

SUMMARY:
The aim of this study was to establish a registration and monitoring system for hypertension in Xinjiang from 2020 to 2030 to obtain real information about patient basic information, patient characteristics, diagnostic test patterns, treatment options, and hospitalization outcomes (including mortality). Treatment complications, hospitalization costs, and end-of-life events (death, major adverse cardiac events, mild adverse cardiovascular events) in patients with hypertension in Xinjiang; and scientific prevention strategies aimed at effectively preventing the onset of hypertension; Guidelines in clinical practice recommend, analyze and develop effective treatment strategies to optimize management and outcomes for patients with hypertension; and create cost-effective assessment systems.

DETAILED DESCRIPTION:
The aim of the study is to establish a platform for monitoring, clinical research and translational medicine in Xinjiang, which aims to provide a basis for future quality improvement and research, and to promote efforts to improve the prognosis of patients with hypertension, and to translate research into improved care for patients, thereby reducing Morbidity and mortality associated with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* A patient diagnosed with primary hypertension who was admitted to the First Affiliated Hospital of Xinjiang Medical University

Exclusion Criteria:

* Patients with secondary hypertension, patients with liver and kidney dysfunction,
* patients with mental disorders, and patients who are unwilling to participate in this trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A patient diagnosed with primary hypertension who was admitted to the First Affiliated Hospital of Xinjiang Medical University
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Resistant hypertension | 10 years of follow-up Resistant hypertension occurred during this period
Death (all-cause mortality, mortality from hypertension complications) | 10 years of follow-up deaths occurred during this period

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 10 years of follow-up deaths occurred during this period

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinjiang Medicial University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No